CLINICAL TRIAL: NCT07163715
Title: Prospective Cohort Study on the Incidence and Associated Factors of Decline in Activities of Daily Living Among Older Adults Discharged From the Emergency Department After a Fall
Brief Title: Incidence and Factors of Functional Decline After Emergency Department Discharge in Older Adults With Falls
Acronym: FALL-ADL
Status: Not yet recruiting | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozge Can. MD, MD, Ege University
Other Study IDs: 25-8T/108
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Fall; Daily Activities; Functional Decline; Older Adults (65 Years and Older)
Keywords: Falls; Decline fictional status; Decline daily activities; Emergency medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this observational study is to learn about changes in activities of daily living (ADL) in older adults after being discharged from the emergency department (ED) following a fall.

The main questions this study aims to answer are:

How often do older adults experience a decline in their ability to perform daily activities after being discharged from the ED for a fall? What health or lifestyle factors (such as frailty, medications, physical activity, or fear of falling) are related to this decline? Participants will be 65 years or older, admitted to the ED for a simple fall, and discharged without hospitalization. At the time of their ED visit, participants will be asked questions about their health, medications, activity level, and daily functioning. They will then be contacted online or by phone at 7 days and 30 days after discharge to answer follow-up questions.

This study will help identify how common functional decline is after falls in older adults discharged from the ED, and which factors may predict higher risk. These findings could help improve follow-up care and prevention strategies for older patients.

DETAILED DESCRIPTION:
Falls are one of the leading causes of morbidity and functional decline in older adults. Even in cases without major injury requiring hospitalization, falls can lead to decreased independence and reduced quality of life. Functional decline, often measured as deterioration in activities of daily living (ADL), is associated with frailty, multimorbidity, polypharmacy, fear of falling, and reduced physical activity. Early identification of older patients at risk for functional decline after an emergency department (ED) visit is critical for designing timely interventions and improving patient outcomes.

This prospective cohort study will enroll 280 patients aged 65 years and older who present to the ED with a simple fall and are discharged without hospitalization. Baseline data will be collected at the time of ED visit, including demographic characteristics, comorbidities, medication use, frailty status (Clinical Frailty Scale), physical activity level (Physical Activity Scale for the Elderly, PASE), fall risk (MEFRAT), and fear of falling (Falls Efficacy Scale-International, FES-I). ADL status will be assessed at baseline and re-assessed at 7 and 30 days after discharge through online or telephone interviews.

The primary outcome is the incidence of decline in ADL within 30 days after ED discharge. Secondary analyses will examine associations between demographic, clinical, functional, and psychosocial factors and the risk of ADL decline, using logistic regression models.

The study is expected to provide valuable insights into the frequency and determinants of functional decline among older adults after ED discharge for falls. Identifying these risk factors will inform strategies for early recognition, follow-up care, and targeted interventions aimed at preventing functional decline and maintaining independence in older patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Presentation to the emergency department with a simple (non-injurious) fall
* Discharged from the ED without hospitalization
* Cognitively able to answer online or telephone follow-up interviews

Exclusion Criteria:

* Falls due to traumatic events other than simple falls
* Hospital admission required after the fall
* Presence of acute confusion, dementia, or other severe cognitive impairment
* Inability to access online or telephone follow-up during the 30-day study period

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: The study population will consist of community-dwelling older adults aged 65 years and older who present to the emergency department (ED) with a simple fall and are discharged without hospitalization. Participants must be cognitively able to complete baseline and follow-up assessments.
  This population represents a group at risk of functional decline despite not requiring inpatient admission. By focusing on older adults discharged from the ED, the study aims to capture real-world outcomes in a population that is often underrepresented in research but commonly experiences falls and subsequent declines in independence.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Decline in Activities of Daily Living | Baseline (ED discharge), 7 days, and 30 days after discharge
  Change in Activities of Daily Living (ADL) score from baseline to follow-up. Decline is defined as an increase in dependency in at least one ADL item compared with baseline.

IPD SHARING:
Plan to Share IPD: No